CLINICAL TRIAL: NCT03776903
Title: Evaluation of the Clinical Performance of the ZIKV Detect™ 2.0 IgM Capture ELISA
Status: Completed | Type: Observational
Sponsor: InBios International, Inc. (Industry)
Collaborators: Fast-Track Drugs & Biologics, LLC (Unknown); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ZIKV-2016-01
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Zika Virus Infection
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endemic: Samples collected from areas endemic for zika. Subject specimens underwent testing with the study device and reference method.
  Interventions: Other: ZIKV Detect™ 2.0 IgM Capture ELISA
- non-endemic: Samples collected from areas non-endemic for zika. Subject specimens underwent testing with the study device and reference method.
  Interventions: Other: ZIKV Detect™ 2.0 IgM Capture ELISA

INTERVENTIONS:
Other: ZIKV Detect™ 2.0 IgM Capture ELISA — De-identified archive specimens are tested by ELISA and compared to reference testing (RT-PCR and CDC MAC-ELISA)

SUMMARY:
The purpose of this study is to evaluate the performance of the ZIKV Detect™ 2.0 IgM Capture ELISA using archived confirmed ZIKV positive and confirmed ZIKV negative human serum samples.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the performance of the ZIKV Detect™ 2.0 IgM Capture ELISA using archived confirmed ZIKV positive and confirmed ZIKV negative human serum samples. The FDA guidance document (ZIKA SEROLOGY DE NOVO/510(K) PRE-MARKET SUBMISSIONS - Recommended Analytical and Clinical Studies for Zika Virus IgM Assays; Dated 02Jun2017; FDA/CDRH/OIR/DMD) allows for the utilization of archival serum specimens to evaluate test performance. This study will follow this guidance. Test samples will be collected from endemic sites (both presumed positive and presumed negative samples) and from non-endemic sites (presumed negative samples). All samples will be shipped to the sponsor for randomization and will be tested at three sites in the United States.

ELIGIBILITY:
Inclusion criteria:

* Human males and females of varying ages and geographical locations where Zika virus is endemic and not endemic.
* Retrospective (archived) and prospective human serum samples. Archived samples will fall under the category of "leftover" specimens as described by FDA guidance.

Exclusion criteria:

• Samples that are not de-identified.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Human males and females of varying ages and geographical locations where Zika virus is endemic and not endemic.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Positive Percent Agreement and Negative Percent Agreement | From symptom onset to 12 weeks after symptom onset.
  The positive percent agreement (PPA) and negative percent agreement (NPA) of the ZIKV Detect™ 2.0 IgM Capture ELISA versus the reference test.

SECONDARY OUTCOMES:
Duration of Positive Percent Agreement | From symptom onset to 12 weeks after symptom onset.
  The time period relative to onset of symptoms that a positive result can be identified and the time period after onset of symptoms that the positive percent agreement is maximized and the longest elapsed time after symptom onset that positive test results are observed.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chu, PhD, Study Director — InBios International
Locations (1):
- InBios International, Seattle, Washington, United States